CLINICAL TRIAL: NCT01709435
Title: A Phase 1 Study of XL184 (Cabozantinib) in Children and Adolescents With Recurrent or Refractory Solid Tumors, Including CNS Tumors
Brief Title: Cabozantinib S-Malate in Treating Younger Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01890; NCI-2012-01890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P121149; COG-ADVL1211; NCI-2013-01571; CDR0000741914; ADVL1211 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1211 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Malignant Solid Neoplasm; Recurrent Melanoma; Recurrent Primary Central Nervous System Neoplasm; Recurrent Thyroid Gland Carcinoma; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Melanoma; Central Nervous System Neoplasms; Thyroid Neoplasms; Carcinoma, Medullary | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cabozantinib S-malate) (Experimental): Patients receive cabozantinib S-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of cabozantinib S-malate in treating younger patients with solid tumors that have come back or no longer respond to treatment. Cabozantinib S-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of XL184 (cabozantinib) (cabozantinib S-malate) administered orally to children with refractory solid tumors including central nervous system (CNS) tumors.

II. To define and describe the toxicities of XL184 (cabozantinib) administered on this schedule.

III. To characterize the pharmacokinetics of XL184 (cabozantinib) in children with refractory solid tumors.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of XL184 (cabozantinib) within the confines of a phase 1 study.

II. To assess the biologic activity of XL184 (cabozantinib). III. To assess the biomarker response (carcinoembryonic antigen [CEA] and calcitonin) in patients with medullary thyroid cancer treated with XL184.

IV. To evaluate overall survival from study entry through a five-year follow-up period.

OUTLINE: This is a dose-escalation study. (Complete as of 4/16/2014)

Patients receive cabozantinib S-malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 6 months, and then annually for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area >= 0.44 m^2 when enrolling on dose level -1; patients must have a body surface area >= 0.35 m^2 when enrolling on dose level 1, 2, or 3
* PART A: Patients with relapsed or refractory solid tumors (excluding medullary thyroid cancer) including CNS tumors and malignant melanoma are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Part B: Patients with medullary thyroid cancer (MTC), with or without bone marrow involvement, will be eligible for Part B; these patients will be enrolled at dose level 2, the recommended phase 2 dose determined in the dose escalation part of the study
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age

  * Note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy:

  * Myelosuppressive chemotherapy: at least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Biologic (anti-neoplastic agent): at least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: at least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * Radiation therapy (XRT): at least 14 days after local palliative XRT (small port); at least 150 days must have elapsed if prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
  * Stem cell infusion without TBI: no evidence of active graft versus (vs.) host disease and at least 56 days must have elapsed after transplant or stem cell infusion
* For patients with solid tumors without known bone marrow involvement:
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients with a solid tumor must be evaluable for hematologic toxicity in the dose-escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male), 1.4 mg/dL (female)
* Urine protein: =< 30 mg/dl in urinalysis or =< 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hour (h) urine sample
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2.8 g/dL
* Prothrombin time (PT) and international normalized ratio (INR) =< 1.5 x ULN
* Serum amylase =< 1.5 x ULN
* Serum lipase =< 1.5 x ULN
* A blood pressure (BP) =< the 95th percentile for age, height, and gender, and not receiving medication for treatment of hypertension; please note that 3 serial blood pressures should be obtained and averaged to determine baseline BP
* Central nervous system function defined as: patients with seizure disorder may be enrolled if receiving non-enzyme inducing anticonvulsants and well controlled
* No history of congenital prolonged corrected QT interval (QTc) syndrome, New York Heart Association (NYHA) class III or IV congestive heart failure (CHF)
* No clinically significant cardiac arrhythmias, stroke or myocardial infarction within 6 months prior to enrollment
* QTc =< 480 msec; Note: patients with grade 1 prolonged QTc (450-480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e. electrolytes, medications)
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Archival tumor tissue slides from either initial diagnosis or relapse must be sent; if tumor tissue is unavailable, the study chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use two methods of birth control - a medically accepted barrier method of contraceptive method (e.g., male or female condom) and a second effective contraceptive method of birth control - during protocol therapy and for at least 4 months after the last dose of XL184; abstinence is an acceptable method of birth control
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients must not be receiving any of the following potent cytochrome P450 family 3, subfamily A, polypeptide 4 cytochrome (CYP3A4) inducers or inhibitors: erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice or St. John's wort
* Patients who are receiving systemic treatment anticoagulation are not eligible; patients receiving prophylactic systemic anticoagulation will be allowed as long as eligibility PT/INR requirements are met
* Patients must not have received enzyme-inducing anticonvulsants within 14 days prior to enrollment
* Patients who are receiving drugs that prolong QTc are not eligible
* Patients must be able to swallow intact tablets; patients who cannot swallow intact tablets are not eligible
* Patients with active bleeding are not eligible; specifically, no clinically significant gastrointestinal (GI) bleeding, GI perforation, intra-abdominal abscess or fistula for 6 months prior to enrollment, no hemoptysis or other signs of pulmonary hemorrhage for 3 months prior to enrollment
* Patients with evidence of an acute intracranial or intratumoral hemorrhage on computed tomography (CT) or magnetic resonance imaging (MRI) are not eligible (patients with evidence of resolving hemorrhage will be eligible)
* Patients who have had or are planning to have the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment
  * Central line placement or subcutaneous port placement is not considered major surgery but must be placed at least 3 days prior to enrollment for external lines (e.g. Hickman or Broviac) and at least 7 days prior to enrollment for subcutaneous port
  * Core biopsy within 7 days prior to enrollment
  * Fine needle aspirate within 7 days prior to enrollment
  * Surgical or other wounds must be adequately healed prior to enrollment
* Patients on antihypertensive therapy for control of blood pressure at the time of enrollment are not eligible
* Patients with any medical or surgical conditions that would interfere with gastrointestinal absorption of this oral agent are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith K Chuk, Principal Investigator — COG Phase I Consortium
Locations (23):
- United States (22):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Dose Level 1: 30 mg/m^2: Patients receive 30 mg/m^2 cabozantinib S-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Part A Dose Level 2: 40 mg/m^2; Part B Dose Level 2: 40 mg/m^2; Part PK Dose Level 2: 40 mg/m^2: Patients receive 40 mg/m^2 cabozantinib S-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Part A Dose Level 3: 55 mg/m^2; Part PK Dose Level 3: 55 mg/m^2: Patients receive 55 mg/m^2 cabozantinib S-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Started | 6 | 9 | 6 | 4 | 10 | 6
Completed | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 6 | 9 | 6 | 3 | 10 | 6
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 5 | 7 | 2 | 2 | 6 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2 | Total
Number analyzed (Participants) | 6 | 9 | 6 | 4 | 10 | 6 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 9 | 6 | 4 | 10 | 6 | 41
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 15.5 [11.0 to 18.0] | 14 [4.0 to 18.0] | 15 [11.0 to 18.0] | 15 [13.0 to 17.0] | 8.5 [5.0 to 17.0] | 10.5 [6.0 to 15.0] | 13 [4.0 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 3 | 2 | 2 | 4 | 20
  Male | 4 | 2 | 3 | 2 | 8 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 9 | 6 | 4 | 10 | 5 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 0 | 2 | 1 | 7
  White | 3 | 6 | 4 | 3 | 5 | 5 | 26
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose of Cabozantinib S-malate
Description: Maximum dose at which fewer than one-third of toxicity-evaluable patients experience a dose limiting toxicity during cycle 1 of therapy.
Time Frame: Up to 28 days
Population: Eligible Patients
Measure: Number; unit: mg/m^2
Arm/Group | Treatment (Cabozantinib S-malate)
Number analyzed (Participants) | 41
mg/m^2 | 40

2. Primary Outcome: Number of Evaluable Patients With Dose Limiting Toxicities of Cabozantinib
Description: Number of toxicity-evaluable patients who experience a dose limiting toxicity during cycle 1 of therapy stratified by dose level and study part.
Time Frame: Up to 28 days
Population: toxicity-evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Number analyzed (Participants) | 6 | 9 | 6 | 4 | 10 | 6
Participants | 0 | 0 | 1 | 1 | 4 | 2

3. Primary Outcome: Clearance of Cabozantinib S-malate
Description: Median (min, max) clearance of cabozantinib stratified by dose level and study part post-dose in cycle 1, day 1.
Time Frame: Up to 24 hours
Population: Eligible Patients
Measure: Median (Full Range); unit: ml/hr
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Number analyzed (Participants) | 6 | 9 | 6 | 4 | 10 | 6
ml/hr | 1641.7 [1020.4 to 2222.2] | 1724.1 [1120.4 to 4477.6] | 3013.8 [1556.4 to 4366.8] | 2281.4 [2247.2 to 2461.5] | 2668.6 [1252.6 to 4801.9] | 1363.8 [1327.4 to 1486.4]

4. Secondary Outcome: Disease Response of Cabozantinib S-malate
Description: Number of response-evaluable patients with response (CR or PR) determined by RECIST guideline (version 1.1) including CR: disappearance of all target and non-target lesions; PR: at least 30% decrease in sum of diameters of target lesions.
Time Frame: Up to 5 years
Population: response-evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Number analyzed (Participants) | 6 | 8 | 6 | 4 | 9 | 6
Participants | 0 | 0 | 1 | 2 | 0 | 1

5. Secondary Outcome: Overall Survival (OS) of Cabozantinib S-malate
Description: Median (95% CI) time to death stratified by dose level and study part.
Time Frame: Up to 5 years
Population: Response evaluable Patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Number analyzed (Participants) | 6 | 8 | 6 | 4 | 9 | 6
Days | 576 [48 to 695] | 1034 [1034 to NA] — The upper limit of the 95% CI is not estimable because the upper limit of the 95% confidence bands does not reach 0.50. This occurs in instances when not enough events have occurred to estimate the parameter. | 869 [163 to 1562] | 256 [190 to 321] | 737 [115 to 1617] | 24 [24 to NA] — The upper limit of the 95% CI is not estimable because the upper limit of the 95% confidence bands does not reach 0.50. This occurs in instances when not enough events have occurred to estimate the parameter.

6. Secondary Outcome: Change From Baseline in VEGF-R2 Concentration
Description: Median (Min, Max) of change for VEGF-R2 sample from baseline to the day 21 or 28 stratified by dose level and study part.
Time Frame: Up to 28 days
Population: Toxicity evaluable patients
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
Number analyzed (Participants) | 6 | 8 | 6 | 4 | 9 | 6
pg/ml | -1121.2 [-1561.4 to -64.8] | -2249.7 [-4385.4 to -764.1] | -2087.3 [-3664.6 to -287.8] | -1287.1 [-2192.0 to -702.5] | -1742.2 [-3409.7 to -221.2] | -2519.4 [-4412.9 to -465.4]

7. Secondary Outcome: Biomarker Response (CEA and Calcitonin) in Patients With Medullary Thyroid Cancer Treated With XL184
Description: Number of patients with tumor markers CEA and/or calcitonin 2x ULN at baseline defined as CR (normalization of CEA or calcitonin) or PR (at least 50% decrease in CEA or CTN) at least 4 weeks apart.
Time Frame: Up to 28 days
Population: Includes Medullary Thyroid Cancer (MTC) patients. The original protocol eligibility did not exclude Medullary Thyroid Cancer (MTC) patients from enrolling onto Part A . The exclusion was added with amendment 5A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part B Dose Level 2: 40 mg/m^2
Number analyzed (Participants) | 1 | 4
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Part A Dose Level 1: 30 mg/m^2 | Part A Dose Level 2: 40 mg/m^2 | Part A Dose Level 3: 55 mg/m^2 | Part B Dose Level 2: 40 mg/m^2 | Part PK Dose Level 2: 40 mg/m^2 | Part PK Dose Level 3: 55 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/6 | 1/9 | 3/6 | 2/4 | 7/10 | 3/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/9 | 3/6 | 2/4 | 6/10 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 6/6 | 4/4 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 30 mg/m^2 (N=6) | Part A Dose Level 2: 40 mg/m^2 (N=9) | Part A Dose Level 3: 55 mg/m^2 (N=6) | Part B Dose Level 2: 40 mg/m^2 (N=4) | Part PK Dose Level 2: 40 mg/m^2 (N=10) | Part PK Dose Level 3: 55 mg/m^2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 30 mg/m^2 (N=6) | Part A Dose Level 2: 40 mg/m^2 (N=9) | Part A Dose Level 3: 55 mg/m^2 (N=6) | Part B Dose Level 2: 40 mg/m^2 (N=4) | Part PK Dose Level 2: 40 mg/m^2 (N=10) | Part PK Dose Level 3: 55 mg/m^2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 1 | 2 | 6 | 2
Abducens nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 0
Accessory nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 3 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 6 | 6 | 4 | 9 | 4
Alkaline phosphatase increased (Investigations) | 3 | 3 | 4 | 2 | 3 | 3
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 2 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1 | 6 | 3
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 6 | 6 | 1 | 8 | 6
Anorexia (Metabolism and nutrition disorders) | 3 | 7 | 4 | 3 | 7 | 5
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 2 | 2 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 6 | 2 | 10 | 5
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 3 | 5 | 2
Blood bilirubin increased (Investigations) | 2 | 1 | 1 | 0 | 2 | 2
Blurred vision (Eye disorders) | 0 | 1 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cardiac troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cholesterol high (Investigations) | 1 | 2 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 6 | 3 | 2 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3 | 4 | 1 | 3
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 3 | 1
Delayed puberty (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 5 | 5 | 4 | 6 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2 | 4 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 1 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Edema face (General disorders) | 1 | 0 | 0 | 2 | 1 | 0
Edema limbs (General disorders) | 1 | 1 | 1 | 0 | 3 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0 | 1
Extraocular muscle paresis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 3 | 8 | 5 | 3 | 7 | 4
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 2 | 2 | 3 | 2 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 2 | 2 | 0 | 0 | 3 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 7 | 2 | 3 | 6 | 3
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 2 | 0 | 2 | 2
Hemoglobin increased (Investigations) | 1 | 2 | 0 | 4 | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 6 | 2 | 3 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 3 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 5 | 4 | 3 | 5 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 7 | 3 | 1 | 6 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 5 | 5 | 3 | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 3 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 1 | 4 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1 | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5 | 3 | 2 | 5 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 6 | 1 | 1 | 6 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 4 | 6 | 5 | 4 | 7 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0
IVth nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 1 | 0 | 3 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1 | 0
Irritability (General disorders) | 0 | 1 | 1 | 0 | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 3 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 3 | 3 | 2 | 3 | 2
Localized edema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 6 | 4 | 3 | 4 | 3
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 3 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 5 | 4 | 4 | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 2 | 3 | 1 | 4 | 3
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 0 | 1 | 3
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 1 | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 2 | 4 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 3 | 2 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pancreatic enzymes decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Penile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 5 | 2 | 4 | 6 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 3 | 7 | 5 | 2 | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 5 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Serum amylase increased (Investigations) | 0 | 1 | 2 | 1 | 2 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 4 | 1 | 2 | 4 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 2 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0 | 2 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 3 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 2 | 2 | 3
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vagus nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 4 | 4 | 7 | 3
Vulval infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 2 | 4 | 5 | 3 | 4 | 3
White blood cell decreased (Investigations) | 6 | 4 | 4 | 1 | 5 | 3
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT01709435/Prot_SAP_000.pdf